CLINICAL TRIAL: NCT00083616
Title: A Phase 2 Multicenter Single Arm Clinical Trial of ABX-EGF Monotherapy in Subjects With Metastatic Colorectal Cancer Following Treatment With Fluoropyrimidine, Irinotecan, and Oxaliplatin Chemotherapy
Brief Title: Evaluating Panitumumab (ABX-EGF) Monotherapy in Patients With Metastatic Colorectal Cancer Following Treatment With Fluoropyrimidine, Irinotecan, and Oxaliplatin Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20030167; NCT00087243 (obsolete NCT alias)
Record Dates: First submitted 2004-05-26; First posted 2004-05-28 (Estimated); Results first posted 2011-07-29 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2013-12

CONDITIONS: Colorectal Cancer; Metastatic Cancer
Keywords: EGFr; Clinical Trial; Panitumumab; ABX-EGF; Immunex; Metastatic Cancer; Vectibix; Abgenix; Amgen
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Panitumumab (Experimental): Participants received panitumumab 6 mg/kg once every 2 weeks weeks administered by intravenous (IV) infusion until progressive disease, inability to tolerate the investigational product, or discontinuation of treatment for other reasons.
  Interventions: Biological: Panitumumab

INTERVENTIONS:
Biological: Panitumumab — Panitumumab 6 mg/kg every once 2 weeks weeks administered by intravenous (IV) infusion.
  Other Names: ABX-EGF; Vectibix

SUMMARY:
The purpose of this study is to determine that panitumumab will have clinically meaningful anti-tumor activity in patients with metastatic colorectal cancer who have developed progressive disease or relapsed while on or after prior fluoropyrimidine, irinotecan and oxaliplatin chemotherapy.

DETAILED DESCRIPTION:
Panitumumab was administered once every 2 weeks until participants developed progressive disease, were unable to tolerate panitumumab, or discontinued treatment for other reasons (eg, administrative decision). Participants then attended a safety follow-up visit 4 weeks from the last panitumumab infusion. Participants were subsequently contacted every 3 months from the last panitumumab infusion through month 24 to assess disease status and survival.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic diagnosis of colorectal adenocarcinoma (diagnostic tissue obtained by tissue biopsy)
* Metastatic colorectal carcinoma
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
* Documented evidence of disease progression during, or following treatment, with fluoropyrimidine, irinotecan and oxaliplatin chemotherapy for metastatic colorectal cancer
* Radiographic documentation of disease progression during or within 6 months following the most recent chemotherapy regimen is required
* Bidimensionally measurable disease
* Tumor expressing epidermal growth factor receptor (EGFr) by immunohistochemistry
* At least 2 but no more than 3 prior chemotherapy regimens for metastatic colorectal cancer
* Adequate hematologic, renal and hepatic function

Exclusion Criteria:

* Symptomatic brain metastases requiring treatment
* Patient with a history of interstitial pneumonitis or pulmonary fibrosis or evidence of interstitial pneumonitis or pulmonary fibrosis
* Use of systemic chemotherapy or radiotherapy within 30 days before enrollment
* Prior epidermal growth factor receptor targeting agents
* Prior anti-tumor therapies including prior experimental agents or approved anti-tumor small molecules and biologics of short (less than 1 week) serum half-life within 30 days before enrollment, or prior experimental or approved proteins with longer serum half-life (e.g., AvastinTM) within 6 weeks before enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2004-03; Primary Completion 2007-05 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Derived] Liao MZ, Prenen H, Dutta S, Upreti VV. The impact of hepatic and renal function on panitumumab exposures in patients with metastatic RAS wild-type colorectal cancer. Cancer Chemother Pharmacol. 2021 Oct;88(4):665-672. doi: 10.1007/s00280-021-04319-w. Epub 2021 Jul 2. PMID 34213592
- See also: FDA-approved Drug Labeling — http://www.vectibix.com/
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 1 March 2004 through 19 Jul 2006. Patient disposition is reported up until the data cut-off date of 22 December 2006. Completed study is defined as participants who either died on study or completed the safety follow-up visit (30 days after the last dose of panitumumab).
Groups:
- Panitumumab (ABX-EGF): Open-label panitumumab administered by intravenous (IV) infusion at a dose of 6 mg/kg given once every 2 weeks until participants developed progressive disease, were unable to tolerate panitumumab, or discontinued treatment for other reasons.
Period: Overall Study
Arm/Group | Panitumumab (ABX-EGF)
Started | 185
Received Study Medication | 182
Completed | 154 (Completed safety followup or died on study as of the data cut-off date of 22 December 2006)
Not Completed | 31
Not completed — Disease Progression | 16
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 3
Not completed — Ineligibility determined | 2
Not completed — Non-compliance | 1
Not completed — Other | 6

BASELINE CHARACTERISTICS:
Groups:
- Panitumumab: Open-label panitumumab administered by intravenous (IV) infusion at a dose of 6 mg/kg given once every 2 weeks until participants developed progressive disease, were unable to tolerate panitumumab, or discontinued treatment for other reasons.
Arm/Group | Panitumumab
Number analyzed (Participants) | 185
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.6 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85
  Male | 100
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Black or African American | 15
  Hispanic or Latino | 19
  Japanese | 0
  Native Hawaiian or Other Pacific Islander | 1
  White or Caucasian | 144
  Other | 2
  Aborigine | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Objective Tumor Response Through Week 16
Description: Confirmed objective tumor response (complete or partial response) based on modified World Health Organization (WHO) criteria, through week 16. Tumor response was assessed by a central Independent Review Committee (IRC) and confirmation 4 weeks after initial assessment was required. Complete Response (CR): Disappearance of all index and non-index lesions and no new lesions. Partial Response (PR): At least a 50% decrease in the sum of the product of the longest diameters (SPD) of index lesions taking as reference the Baseline SPD, and no new non-index lesions and no "unequivocal progression" of non-index lesions, or, the disappearance of all index lesions and persistence of one or more non-index lesions not qualifying for either CR or Progressive Disease.
Time Frame: 16 weeks
Population: Adjudicated Prior Failures Set, composed of participants confirmed to be eligible by the Independent Eligibility Review Committee (IERC)
Measure: Number; unit: Participants
Arm/Group | Panitumumab
Number analyzed (Participants) | 142
Participants | 5

2. Primary Outcome: Duration of Response
Description: The time from first objective response to first observed progression of disease or death if the death was due to disease progression (whichever comes first); participants who respond and have not progressed while on study or died for reasons other than disease progression while on study were censored at their last evaluable disease assessment date. Response (complete or partial response) was assessed per modified WHO criteria by the central IRC. Complete Response (CR): Disappearance of all index and non-index lesions and no new lesions. Partial Response (PR): At least a 50% decrease in the sum of the product of the longest diameters (SPD) of index lesions taking as reference the Baseline SPD, and no new non-index lesions and no "unequivocal progression" of non-index lesions, or, the disappearance of all index lesions and persistence of one or more non-index lesions not qualifying for either CR or Progressive Disease.
Time Frame: Until the data cut-off date of 22 December 2006. Maximum time of follow-up was 128 weeks.
Population: Subset of the Adjudicated Prior Failures Set, composed of participants confirmed to be eligible by the Independent Eligibility Review Committee (IERC), who had a confirmed obective tumor response
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Panitumumab
Number analyzed (Participants) | 5
Weeks | 14.0 [12.4 to 101.7]

3. Secondary Outcome: Number of Participants With Objective Tumor Response Throughout Study
Description: Confirmed objective tumor response (complete or partial response) based on modified World Health Organization (WHO) criteria, throughout the duration of the study Tumor response was assessed by a central Independent Review Committee (IRC) and confirmation 4 weeks after initial assessment was required. Complete Response (CR): Disappearance of all index and non-index lesions and no new lesions. Partial Response (PR): At least a 50% decrease in the sum of the product of the longest diameters (SPD) of index lesions taking as reference the Baseline SPD, and no new non-index lesions and no "unequivocal progression" of non-index lesions, or, the disappearance of all index lesions and persistence of one or more non-index lesions not qualifying for either CR or Progressive Disease.
Time Frame: Until the data cut-off date of 22 December 2006. Maximum time of follow-up was 128 weeks.
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Panitumumab
Number analyzed (Participants) | 142
Participants | 5

4. Secondary Outcome: Time to Response
Description: Median time from enrollment to objective tumor response for participants who responded.
Time Frame: Until the data cut-off date of 22 December 2006. Maximum time of follow-up was 128 weeks.
Population: Subset of Adjudicated Prior Failures Set, composed of participants confirmed to be eligible by the Independent Eligibility Review Committee (IERC), who had a confirmed objective tumor response
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | Panitumumab
Number analyzed (Participants) | 5
Weeks | 11.0 [7.7 to 11.1]

5. Secondary Outcome: Progression-free Survival Time
Description: Kaplan-Meier estimate of median time from enrollment to death or first observed disease progression (whichever comes first). Participants who did not progress while on study and did not die while on study were censored at the last evaluable disease assessment date.
Time Frame: Until the data cut-off date of 22 December 2006. Maximum follow-up time was 128 weeks.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Panitumumab
Number analyzed (Participants) | 142
Weeks | 7.3 [7.1 to 7.4]

6. Secondary Outcome: Time to Disease Progression
Description: Kaplan-Meier estimate of the median time from enrollment to first observed disease progression or death if death was due to disease progression (whichever comes first). Participants who did not progress while on study or died for reasons other than disease progression while on study were censored at their last evaluable disease assessment date.
Time Frame: Until the data cut-off date of 22 December 2006. Maximum follow-up time was 128 weeks.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Panitumumab
Number analyzed (Participants) | 142
Weeks | 7.3 [7.1 to 7.6]

7. Secondary Outcome: Time to Treatment Failure
Description: Kaplan-Meier estimate of median time from enrollment to treatment failure, defined as the date the decision was made to end treatment. Participants remaining in the treatment phase at the time of the analysis were censored on their last visit date.
Time Frame: Until the data cut-off date of 22 December 2006. Maximum follow-up time was 128 weeks.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Panitumumab
Number analyzed (Participants) | 142
Weeks | 8.0 [7.4 to 8.1]

8. Secondary Outcome: Duration of Stable Disease
Description: Kaplan-Meier estimates of the median time from enrollment to the date of first observed disease progression or death due to disease progression among those participants with a best outcome of stable disease. Stable disease (SD): Neither sufficient shrinkage of Index lesions to qualify for partial response nor sufficient increase to qualify for progressive disease (PD) taking as reference the nadir sum of the products of the longest diameters (SPD) since the treatment started and the disappearance of or persistence of one or more non-index lesions not qualifying for PD.
Time Frame: Until the data cut-off date of 22 December 2006. Maximum follow-up time was 128 weeks.
Population: Subset of Adjudicated Prior Failures Set, composed of participants confirmed to be eligible by the Independent Eligibility Review Committee (IERC), with a best outcome of stable disease
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Panitumumab
Number analyzed (Participants) | 31
Weeks | 23.9 [23.0 to 31.0]

9. Secondary Outcome: Overall Survival
Description: Kaplan-Meier estimate of median time from enrollment to death from any cause. Deaths were recorded during treatment, safety follow-up and long term follow-up.
Time Frame: Until the data cut-off date of 22 December 2006. Maximum follow-up time was 128 weeks.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Panitumumab
Number analyzed (Participants) | 142
months | 7.0 [5.7 to 8.0]

ADVERSE EVENTS:
Time Frame: From the first dose through maximum of safety follow-up or 30 days after last dose; maximum time on study treatment was 1.25 years.
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
Arm/Group | Panitumumab
Serious Adverse Events (participants affected / at risk) | 62/182
Other Adverse Events (participants affected / at risk) | 176/182
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Panitumumab (N=182)
Anaemia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 3
Abdominal hernia (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 4
Abdominal pain lower (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 3
Colonic fistula (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Duodenal obstruction (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Pancreatitis (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Reflux oesophagitis (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 2
Early satiety (General disorders) | 1
Fatigue (General disorders) | 1
Pain (General disorders) | 1
Bile duct obstruction (Hepatobiliary disorders) | 2
Cholangitis (Hepatobiliary disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Jaundice cholestatic (Hepatobiliary disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Bacteraemia (Infections and infestations) | 1
Catheter related infection (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Endocarditis staphylococcal (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Lobar pneumonia (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 3
Pneumonia bacterial (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Septic embolus (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1
Weight decreased (Investigations) | 1
Cachexia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1
Fluid retention (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Anoxic encephalopathy (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 1
Hepatic encephalopathy (Nervous system disorders) | 1
Speech disorder (Nervous system disorders) | 1
Spinal cord compression (Nervous system disorders) | 1
Vocal cord paralysis (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 2
Confusional state (Psychiatric disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4
Circulatory collapse (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 3
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Panitumumab (N=182)
Abdominal pain (Gastrointestinal disorders) | 34
Ascites (Gastrointestinal disorders) | 11
Constipation (Gastrointestinal disorders) | 36
Diarrhoea (Gastrointestinal disorders) | 48
Dyspepsia (Gastrointestinal disorders) | 12
Nausea (Gastrointestinal disorders) | 58
Stomatitis (Gastrointestinal disorders) | 16
Vomiting (Gastrointestinal disorders) | 38
Asthenia (General disorders) | 12
Chills (General disorders) | 11
Fatigue (General disorders) | 66
Oedema peripheral (General disorders) | 17
Pyrexia (General disorders) | 23
Paronychia (Infections and infestations) | 32
Rash pustular (Infections and infestations) | 16
Urinary tract infection (Infections and infestations) | 13
Weight decreased (Investigations) | 19
Anorexia (Metabolism and nutrition disorders) | 31
Decreased appetite (Metabolism and nutrition disorders) | 11
Dehydration (Metabolism and nutrition disorders) | 12
Hypokalaemia (Metabolism and nutrition disorders) | 15
Hypomagnesaemia (Metabolism and nutrition disorders) | 20
Back pain (Musculoskeletal and connective tissue disorders) | 21
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10
Dizziness (Nervous system disorders) | 12
Headache (Nervous system disorders) | 18
Anxiety (Psychiatric disorders) | 14
Depression (Psychiatric disorders) | 10
Insomnia (Psychiatric disorders) | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 24
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 29
Acne (Skin and subcutaneous tissue disorders) | 10
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 125
Dry skin (Skin and subcutaneous tissue disorders) | 28
Erythema (Skin and subcutaneous tissue disorders) | 112
Exfoliative rash (Skin and subcutaneous tissue disorders) | 30
Nail disorder (Skin and subcutaneous tissue disorders) | 15
Pruritus (Skin and subcutaneous tissue disorders) | 96
Rash (Skin and subcutaneous tissue disorders) | 44
Rash papular (Skin and subcutaneous tissue disorders) | 12
Skin exfoliation (Skin and subcutaneous tissue disorders) | 17
Skin fissures (Skin and subcutaneous tissue disorders) | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.